CLINICAL TRIAL: NCT00758147
Title: Assessment of Force Feedback Joystick in Upper Limb Rehabilitation Following Stroke
Brief Title: Force Feedback Joystick in Upper Limb Rehabilitation Following Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Ono Academic College (Other)
Responsible Party: Shai Brill M.D, Beit Rivka Geriatric Center
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BGC085012CTIL
Record Dates: First submitted 2008-09-21; First posted 2008-09-23 (Estimated); Last update posted 2008-09-23 (Estimated); Status verified 2008-09

CONDITIONS: Stroke
Keywords: force feedback joystick; stroke; haptics; kinematics; rehabilitation; robotics; Force feedback joystick in stroke rehabilitation
MeSH Terms: conditions — Stroke | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Exercise with force feedback joystick — System consists of a commercially available force feedback joystick, and specially written software. Patients will work with the system 5 times a week for 4 weeks, a half hour each time, 2 weeks with visual and haptic feedback and 2 weeks without the feedback.

SUMMARY:
The purpose of this study is to assess the influence of force feedback joysticks and haptic feedback in improving upper limb rehabilitation outcomes following stroke.

DETAILED DESCRIPTION:
Upper limb paresis or plegia following stroke remains a significant cause of impairment and disability. Regaining function requires learning through repetitive movements and activities of daily living(ADLs).

The aim of the study in this application is to test the usability of the system in specialized rehabilitation hospital settings. In this first stage of development, after developing and testing the system together with expert physiotherapists, we will examine the system for usability (is it "user friendly"), comfort level, and therapeutic efficacy.

The system consists of an ordinary PC computer, specially written software, and a commercially available force feedback joystick. (Force feedback joysticks, are usually used for gaming; they contain miniature motors that allow the joystick to either help or resist the movements of the person using it). Patients who are unable to grasp the joystick will use a specially built arm rest that is attached to an ordinary office chair without wheels. Patients rest their forearm on the arm rest and thus can manipulate the joystick by means of movement of the shoulder and elbow joints instead of by movements of the wrist, since wrist movements are often difficult for brain damaged individuals.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable post first stroke patients
* Score of more than 17 on the Mini Mental Scale Test(MMST)

Exclusion Criteria:

* A history of psychiatric illness
* Inability to understand the informed consent form
* Inability to understand and follow 2-3 step instructions
* Receptive aphasia (sensory aphasia)

Ages: 65 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-11 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer impairment scale | 1 month
Wolf Motor Function Test | One month

SECONDARY OUTCOMES:
Satisfaction survey about the use of the joystick | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Shai Brill, M.D., Principal Investigator — Beit Rivka Geriatric Hospital; Heidi Sugarman, PhD, Study Director — Ono Academic College
Locations (1):
- Beit Rivka Geriatric Hospital, Petah Tikva, Israel